CLINICAL TRIAL: NCT01541501
Title: Phase 4 Study of Comparison Among 3 Different No-contact Instruments to Valuate Central Corneal Thickness
Brief Title: Comparison of Three Different No-contact Pachymetries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luigi Varano, MD - Principal Investigator, M. D., University of Catanzaro
Other Study IDs: PAK-NC
Record Dates: First submitted 2012-02-20; First posted 2012-03-01 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Corneal Thickness
Keywords: Central Corneal Thickness; Pachymetry
MeSH Terms: interventions — Corneal Pachymetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pachymetry: All recruited volunteers in present study, that underwent pachymetry measurement with four different instruments
  Interventions: Device: Pachymetry

INTERVENTIONS:
Device: Pachymetry — Healthy volunteers recruited among subject that underwent a routine ophthalmologic evaluation or among both students and workers at our clinic, will be submitted to CCT measurement through four different instruments: Scheimpflug camera tomography, SD-OCT, anterior chamber SD-OCT, and finally with US pachymeter.
  Other Names: Scheimpflug camera tomography (Pentacam© HR - Oculus ind., Wetzlar, Germany).; SD-OCT (RTVue© - Optovue inc. Fremont, CA, USA).; anterior chamber SD-OCT (CASIA©, Tomey corp., Nagoya, Japan).; Ultrasound pachymeter (Pacline© - Optikon ind., Rome, Italy).

SUMMARY:
Study wants to compare central corneal thickness (CCT) obtained through 3 different no-contact instruments and to compare them with contact ultrasound pachymetry, actually the gold standard technique.

DETAILED DESCRIPTION:
Corneal pachymetry is the measurement of corneal thickness, usually expressed in microns (μ).

Pachymetry is systematically used for the monitoring of corneal oedema, for the management and assessment of the progression risk of the ocular hypertension, for the diagnosis, the management and follow-up of keratoconus, as well as it is important in the pre and postoperative management of corneal surgical procedures. CCT is a factor well known to influence tonometry. Its assessment is fundamental in glaucoma practice to allow a correct intraocular pressure (IOP) evaluation.

The purpose of this study is to compare CCT measurements using four different instruments: Scheimpflug camera tomography, spectral-domain optical coherence tomography (SD-OCT), anterior chamber SD-OCT and ultrasound pachymetry.

ELIGIBILITY:
Inclusion Criteria:

* subjects that gave a valid consensus to be included in this experimentation,
* aged between 18 and 75 years,
* Best-Corrected Visual Acuity (BCVA) of 20/100 or better,
* refraction included between -6 and +6 dioptres,
* astigmatism included between -2 and +2 dioptres.

Exclusion Criteria:

* History of refractive surgery or any keratoplasty procedure,
* corneal opacities or diseases that make not suitable applanation tonometry or pachymetry.
* Use of contact lenses.
* History of corneal dystrophies or degenerative diseases, (like keratoconus and pellucid marginal degeneration).
* History of glaucoma or ocular hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers recruited among subject that underwent a routine ophthalmologic evaluation or among both students and workers at our clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Central Corneal Thickness (CCT) expressed in microns (μm) | partecipants will be followed for one day, i. e. until the CCT measurements with all instruments object of present study are taken
  to valuate differences among all obtained no-contact CCT measurements and compare them with the CCT measured with the reference tool (Ultrasound pachymeter).

SECONDARY OUTCOMES:
Central Corneal Thickness (CCT) expressed in microns (μm) | partecipants will be followed for one day, i. e. until the CCT measurements with all instruments object of present study are taken
  to valuate test-retest reliability of each instrument

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Varano, M. D., Principal Investigator — University of Catanzaro
Locations (1):
- University of Catanzaro - Eye Department, Catanzaro, Italy